CLINICAL TRIAL: NCT06541574
Title: Prevention of ProliFerative Vitreoretinopathy with Intravitreal MethotreXate in Primary Retinal DEtachment Repair (FIXER) Trial
Acronym: FIXER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cincinnati Eye Institute, Southwest Ohio (Other)
Responsible Party: Principal Investigator, Christopher Riemann, Principal Investigator, Cincinnati Eye Institute, Southwest Ohio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIXER-PVR
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Proliferative Vitreoretinopathy; Rhegmatogenous Retinal Detachment
Keywords: Proliferative Vitreoretinopathy; Rhegmatogenous Retinal Detachment
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Methotrexate; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: 1:1:1:1 randomization strategy into four groups:
  1. Control group - receiving no methotrexate
  2. Injection group - receiving standard surgery without intraoperative methotrexate followed by postoperative 400µg intravitreal methotrexate injections 1, 3, 6, and 10 weeks after surgery.
  3. Infusion group - receiving surgery with intraoperative intraocular methotrexate infusion as described above and postoperative sham injections.
  4. Combined Infusion/Injection group - receiving both intraoperative intraocular methotrexate infusion and postoperative 400µg intravitreal methotrexate injections 1, 3, 6, and 10 weeks after surgery.
Who Masked: Participant, Investigator
Masking Description: The Doctor Administring the medication are not masked and are not involved with primary follow up of the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (Sham Comparator): receiving no methotrexate
  Interventions: Drug: Sham Injection
- Injection group (Experimental): receiving standard surgery without intraoperative methotrexate followed by postoperative 400µg intravitreal methotrexate injections 1, 3, 6, and 10 weeks after surgery.
  Interventions: Drug: Methotrexate Injection
- Infusion Group (Experimental): receiving surgery with intraoperative intraocular methotrexate infusion as described above and postoperative sham injections.
  Interventions: Drug: Methotrexate Infusion
- Combined Infusion/Injection group (Experimental): receiving both intraoperative intraocular methotrexate infusion and postoperative 400µg intravitreal methotrexate injections 1, 3, 6, and 10 weeks after surgery.
  Interventions: Drug: Methotrexate Injection; Drug: Methotrexate Infusion

INTERVENTIONS:
Drug: Methotrexate Injection — Methotrexate injection
  Arms: Combined Infusion/Injection group; Injection group
Drug: Methotrexate Infusion — Methotrexate Infusion
  Arms: Combined Infusion/Injection group; Infusion Group
Drug: Sham Injection — Sham Injection
  Arms: Control Group

SUMMARY:
I. Title Prevention of ProliFerative Vitreoretinopathy with Intravitreal MethotreXate in Primary Retinal DEtachment Repair (FIXER) Trial

* Today's Date: September 18, 2023 II. Principal Investigator
* Principal Investigator: Christopher D. Riemann, M.D. (Cincinnati Eye Institute)
* Email: criemann@cvphealth.com, Phone: 513-708-1979

V. Research Summary

Purpose:

To evaluate methotrexate for the prevention of PVR after primary rhegmatogenous retinal detachment repair.

Methods:

Inclusion Criteria:

• Any adult patient, age ≥18 years-old, undergoing primary rhegmatogenous retinal detachment surgery with pars plana vitrectomy at the Cincinnati Eye Institute in Blue Ash, Ohio who is able to give informed consent.

Exclusion Criteria:

* Age <18 years old
* Pregnant patients or patients of child bearing potential unwilling to utilize long term contraception for the 12-week period spanning vitrectomy surgery for retinal detachment repair up until the 3 month postoperative visit.
* History of endophthalmitis, ruptured globe or significant trauma in the affected eye
* Chronic retinal detachment (symptoms greater than or equal to six weeks)
* Any previous previous retinal detachment repair with pars plana vitrectomy, or scleral buckling surgery. Patients having undergone previous pneumatic retinopexy will not be excluded.
* Presence of Grade C PVR: full thickness retinal folds or subretinal bands
* Patients with contraindications to methotrexate, including breastfeeding, pregnancy, attempting to conceive a child or any known hypersensitivity or intolerance to methotrexate
* Patients with diminished mental capacity precluding their ability to give informed consent.

Study Design and Randomization This prospective double masked trial will randomize patients into four groups in a 1:1:1:1 fashion. All attending surgeons and patients will be masked to group randomization. Randomization into four groups will occur on the day of surgery by the Cincinnati Eye Institute's pharmacist, Deepali Chachare. Group A will consist of ≥ 150 patients receiving intraoperative infusion with balanced salt solution containing methotrexate (40mg/500mL BSS), and methotrexate intravitreal injections (400mcg/0.05mL) at postoperative weeks 1, 3, 6, and 10. Group B will consist of ≥ 150 patients receiving intraoperative balanced salt solution infusion containing methotrexate, and sham intravitreal injections at postoperative weeks 1, 3, 6, and 10. Group C will consist of ≥ 150 patients receiving a balanced salt solution infusion without methotrexate, and methotrexate injections at postoperative weeks 1, 3, 6, and 10. Group D will consist of ≥ 150 patients receiving intraoperative balanced salt solution infusion without methotrexate, and sham intravitreal injections at postoperative weeks 1, 3, 6, and 10.

DETAILED DESCRIPTION:
I. Title Prevention of ProliFerative Vitreoretinopathy with Intravitreal MethotreXate in Primary Retinal DEtachment Repair (FIXER) Trial

IV. General Study Information ing on the surgeon and technique, successful retinal reattachment rates range from 70-80% for PR, and even higher with SB and/or PPV.10 Proliferative vitreoretinopathy (PVR), the formation of proliferative fibrocellular membranous tissue overlying the retina, can cause contracture and subsequent recurrent tractional retinal detachment. PVR is the leading cause of failure following RRD repair, complicating 10% of routine RRD procedures and a higher fraction of RRD in the setting of higher risk scenarios and occurs approximately 4,000 times per year in the US.11,12 Risk factors for PVR formation, including duration of RRD, uveitis, myopia (≥ -5.00), lens status, number of retinal breaks, size of breaks, duration of photopsias/floaters/shadows, presence of macula detachment, giant retinal tears, vitreous hemorrhage, and history of trauma. These risk factors will all be collected. Intraoperative data collected will include vitrectomy gauge, use of a drainage retinotomy, use of scleral buckle, type of retinal tamponade (air, SF6, C3F8, or silicone oil), fellow surgeon involvement, duration of surgery, development of choroidal detachment, amount of laser spots, amount of laser energy, number of retinal breaks, total clock hours of retinal breaks, and surgical complications. Surgically removing PVR to reattach the retina can be exceedingly challenging, resulting in poor visual outcomes, with reattachment rates ranging from 60-80%.11 Furthermore, even with successful anatomic reattachment, only 40-80% of patients recover ambulatory vision or better.11 The most commonly cited classification system to grade PVR is the updated Retina Society Classification in 2016. This system describes PVR into grades A-C with increasing severity. Grade A PVR is described as haziness in the vitreous haze or clumps of pigment, representing the migration of RPE cells into the vitreous. Grade B is described wrinkling of the retinal surface, rolled edges of a retinal tear, or retinal stiffness. Grade C-Posterior is described as a full-thickness retinal folds or subretinal strands posterior to equator. Grade C-Anterior is described as full-thickness retinal folds or subretinal strands anterior to equator, anterior displacement, and condensed vitreous strands.13

As of this writing, there are no prospective human studies demonstrating that a prophylactic medication can successfully prevent PVR. PVR prevention represents a significant unmet medical need. Methotrexate's proven antiproliferative and anti-inflammatory properties make it a promising candidate for prevention of PVR. Methotrexate exerts several anti-inflammatory and antiproliferative biochemical mechanisms, including competitive antagonism of dihydrofolate reductase, inhibition of purine and pyrimidine synthesis, transmethylation reactions, and nitric oxide production.14 Moreover, methotrexate has long been used to treat intraocular lymphoma and refractory uveitis, with an established intraocular dosing regimen and excellent intraocular safety profiles as described above.

Based on these long established - now standard of care - protocols in the ocular oncology and uveitis literature, a rational dosing strategy for our study of methotrexate for PBVR prevention was established as follows. The standard intravitreal dose of methotrexate for primary intraocular lymphoma and refractory posterior uveitis is 400mcg into an approximately 5mL eye. Dosing regimens for these two diseases are typically two injections per week for 1 month, 1 injection per week for 2 months and 1 injection per month for 9 additional months. Extensive off-label clinical experience by our group with methotrexate for PVR prevention in high-risk scenarios (going back to 2006) has led our group to believe that this very aggressive dosing regimen is not needed for a substantial anti PVR effect. Furthermore, the well documented side effect of corneal toxicity is much less frequent at a less aggressive dosing regimen and to that end we have adapted the following dosing strategy. During vitrectomy surgery for retinal detachment repair, 40mg of methotrexate is placed into a 500mL bottle of BSS intraocular irrigation solution yielding and identical final intraocular concentration of methotrexate that is equal to a 400mcg injection into a 5 mL eyeball. Methotrexate is a small and readily soluble molecule so an equilibrium of therapeutic tissue concentrations is achieved quickly. Following the aqueous phase of retinal detachment surgery, the (methotrexate containing) BSS infusion is turned off, all intraocular BSS is removed and replaced with a vitreous fill of either air, gas, or silicon oil. The resulting dramatically altered distribution volume of any water-soluble drug makes intraoperative injection dosing at the end of the surgical case very problematic. The intraoperative infusion methodology eliminates these concerns and doses the eye at the time when surgical manipulation and injury (which are felt to be causative factors in PVR formation) occur. We selected the intraoperative intraocular infusion strategy because of the direct and controlled ocular drug delivery, the ease of this dosing strategy, the simplicity of masking both the surgeon and patient (with an opaquer plastic bag covering the infusion bottle), and the elimination of systemic side effect concerns. Our postoperative injection regimen of 400mcg intravitreal injections - one, three, six, and ten weeks postoperatively - was developed to: 1) provide greatest antiproliferative and anti-inflammatory effects closer to the period of surgical injury, 2) maintain persistent effects through the typical PVR formation window of 4 - 8 weeks after surgery, and 3) minimize the corneal toxicity of accumulating methotrexate exposure. Our group has published and presented convincing evidence that both intraoperative infusion and postoperative injection dosing have clinical efficacy. It remains to be elucidated whether the infusion approach, the injection approach or a combination of both are needed for optimal effect. This is the underlying rationale for the 1:1:1:1 randomization strategy into four groups.

Detailed Study Visit Description

The Study will consist of 11 visits spread out over about 12 months. These are summarized in the table attached below. In order:

Visit Number -1 (Preop / screening): 1 - 14 days prior to surgery This is the visit at which the patient's retinal detachment will be diagnosed and the surgical plan for repair established.

Snellen visual acuity and (optional) ETDRS visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. The patient will be screened for inclusion and exclusion criteria Pregnancy screen and contraception discussion as appropriate for patients of child bearing potential The detained geometry of the retinal detachment and associated retinal pathologies will be recorded Recording of PVR risk factors Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy The patient will sign the clinic based informed consent to proceed with surgery.

If the patient meets the inclusion criteria for the trial, the patient will be invited to participate in the trial and be given the study informed consent document to review.

The patient will be tentatively randomized into one of the 4 study groups to aid with preoperative work flow and possible methotrexate preparation requirements for surgery.

Visit Number 0 (Surgery):

The ambulatory surgery center informed consent to treat will be signed Pregnancy screen and contraception discussion as appropriate for patients of child bearing potential The study informed consent document is signed by the patient. The patient will be definitively randomized into one of the 4 study groups. Vitrectomy surgery for retinal detachment repair will be performed The detained geometry of the retinal detachment and associated retinal pathologies will be recorded Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy

Visit Number 1 (Postop Day 1):

Snellen visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects

Visit Number 2 (Postop Week 1) ± 3 days:

Snellen visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects Pregnancy screen and contraception discussion as appropriate for patients of child bearing potential Sham or real methotrexate injection according to patient study group randomization by unmasked investigator

Visit Number 3 (Postop Week 3) ± 3 days:

Snellen visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects Pregnancy screen and contraception discussion as appropriate for patients of child bearing potential Sham or real methotrexate injection according to patient study group randomization by unmasked investigator

Visit Number 4 (Postop Week 6) ± 7 days:

Snellen visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects Pregnancy screen and contraception discussion as appropriate for patients of child bearing potential Sham or real methotrexate injection according to patient study group randomization by unmasked investigator

Visit Number 5 (Postop Week 10) ± 7 days:

Snellen visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects Pregnancy screen and contraception discussion as appropriate for patients of child bearing potential Sham or real methotrexate injection according to patient study group randomization by unmasked investigator

Visit Number 6 (Postop Month 4) ± 14 days:

Snellen visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects

Visit Number 7 (Postop Month 6) ± 28 days:

Snellen visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects

Visit Number 8 (Postop Month 9) ± 28 days:

Snellen visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects

Visit Number 9 (Postop Month 12) ± 28 days:

Snellen visual acuity will be obtained ETDRS visual acuity will be obtained IOP will be determined Slit lamp exam and dilated fundus exam will be performed and recorded. Recording of presence of PVR and or ERM Recording of presence of corneal epitheliopathy Recording of other ocular methotrexate side effects

VI. Statistical Analysis All data will be tabulated on a secure Microsoft Excel document. All information will be stored on a password protected Cincinnati Eye Institute computer on its secure HIPPA compliant network. Only study investigators will have password access to this secure spreadsheet. An Analysis of Variance (ANOVA) table will be generated for each variable to determine statistical significance (p < 0.05).

Statistical power calculations show that an N of 215 patients in each group will allow for detection of a reduction in PVR rate from 10% to 5% and an N of 50 patients will allow for detection of a reduction in PVR rate from 10% to 1% so this study should be fully recruited in approximately 1 year given current patient volumes.

ELIGIBILITY:
Inclusion Criteria:

• Any adult patient, age > 18 years-old, undergoing primary rhegmatogenous retinal detachment surgery with pars plana vitrectomy at the Cincinnati Eye Institute in Blue Ash, Ohio who is able to give informed consent.

Exclusion Criteria:

* Age <18 years-old
* Pregnant patients or patients of child bearing potential unwilling to utilize long term contraception for the 12-week period spanning vitrectomy surgery for retinal detachment repair up until the 3 month postoperative visit.
* History of endophthalmitis, ruptured globe or significant trauma in the affected eye
* Chronic retinal detachment (symptoms > six weeks)
* Any previous previous retinal detachment repair with pars plana vitrectomy, or scleral buckling surgery. Patients having undergone previous pneumatic retinopexy will not be excluded.
* Presence of Grade C PVR: full thickness retinal folds or subretinal bands
* Patients with contraindications to methotrexate, including breastfeeding, pregnancy, attempting to conceive a child or any known hypersensitivity or intolerance to methotrexate
* Patients with diminished mental capacity precluding their ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | Month 12
  Percentage of patients achieving single Surgery Success rate for primary Rhegmatogenous Retinal Detachment repair in each group.

SECONDARY OUTCOMES:
number of retinal detachment repair reoperations | 12 months
  Comparison of number of retinal detachment repair reoperations between study groups
Visual Acuity | 12 months
  Mean final Visual Acuity within and between study groups
Time to Re-detachment from PVR | 12 months
  Time to Re-detachment from PVR
methotrexate-associated corneal epitheliopathy | 12 months
  number of patients developing methotrexate-associated corneal epitheliopathy
Complications | 12 months
  Rate of development of complications (epiretinal membrane formation, endophthalmitis, other ophthalmic surgeries)
Incidence of PVR | 12 months
  Incidence of PVR amongst the study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Eye Institute, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCannel CA. Meta-analysis of endophthalmitis after intravitreal injection of anti-vascular endothelial growth factor agents: causative organisms and possible prevention strategies. Retina. 2011 Apr;31(4):654-61. doi: 10.1097/IAE.0b013e31820a67e4. PMID 21330939
- [Background] Dave VP, Pathengay A, Schwartz SG, Flynn HW Jr. Endophthalmitis following pars plana vitrectomy: a literature review of incidence, causative organisms, and treatment outcomes. Clin Ophthalmol. 2014 Oct 31;8:2183-8. doi: 10.2147/OPTH.S71293. eCollection 2014. PMID 25382968
- [Background] Habot-Wilner Z, Frenkel S, Pe'er J. Efficacy and safety of intravitreal methotrexate for vitreo-retinal lymphoma - 20 years of experience. Br J Haematol. 2021 Jul;194(1):92-100. doi: 10.1111/bjh.17451. Epub 2021 Apr 26. PMID 33900619
- [Background] Choudhury H, Jindal A, Pathengay A, Flynn HW Jr. An outbreak of Ralstonia pickettii endophthalmitis following intravitreal methotrexate injection. Clin Ophthalmol. 2015 Jun 23;9:1117-20. doi: 10.2147/OPTH.S81218. eCollection 2015. PMID 26150690
- [Background] Zhou X, Zhou X, Shi H, Lai J, Wang Q, Li Y, Chen K, Li Q, Zhou Q, Cao X, Chen B, Xiao J. Reduced frequency of Intravitreal methotrexate injection lowers the risk of Keratopathy in Vitreoretinal lymphoma patients. BMC Ophthalmol. 2020 May 12;20(1):189. doi: 10.1186/s12886-020-01464-3. PMID 32397978
- [Background] Sadaka A, Sisk RA, Osher JM, Toygar O, Duncan MK, Riemann CD. Intravitreal methotrexate infusion for proliferative vitreoretinopathy. Clin Ophthalmol. 2016 Sep 19;10:1811-1817. doi: 10.2147/OPTH.S111893. eCollection 2016. PMID 27698550
- [Background] Noble CW, Kim HJ, Pham H, Riemann CD. Prophylactic intravitreal methotrexate for PVR prevention in patients undergoing primary RRD repair with PPV with history of contralateral PVR. American Society of Retina Specialists Annual Meeting. Virtual July 24-26, 2020.
- [Background] Ivanisevic M. The natural history of untreated rhegmatogenous retinal detachment. Ophthalmologica. 1997;211(2):90-2. doi: 10.1159/000310766. PMID 9097312
- [Background] SCHEPENS CL, OKAMURA ID, BROCKHURST RJ. The scleral buckling procedures. I. Surgical techniques and management. AMA Arch Ophthalmol. 1957 Dec;58(6):797-811. doi: 10.1001/archopht.1957.00940010819003. No abstract available. PMID 13478226
- [Background] Steel D. Retinal detachment. BMJ Clin Evid. 2014 Mar 3;2014:0710. PMID 24807890
- [Background] Pastor JC. Proliferative vitreoretinopathy: an overview. Surv Ophthalmol. 1998 Jul-Aug;43(1):3-18. doi: 10.1016/s0039-6257(98)00023-x. PMID 9716190
- [Background] Rachal WF, Burton TC. Changing concepts of failures after retinal detachment surgery. Arch Ophthalmol. 1979 Mar;97(3):480-3. doi: 10.1001/archopht.1979.01020010230008. PMID 420635
- [Background] Di Lauro S, Kadhim MR, Charteris DG, Pastor JC. Classifications for Proliferative Vitreoretinopathy (PVR): An Analysis of Their Use in Publications over the Last 15 Years. J Ophthalmol. 2016;2016:7807596. doi: 10.1155/2016/7807596. Epub 2016 Jun 27. PMID 27429798
- [Background] Chan ES, Cronstein BN. Methotrexate--how does it really work? Nat Rev Rheumatol. 2010 Mar;6(3):175-8. doi: 10.1038/nrrheum.2010.5. PMID 20197777
- [Background] BSS- basic salt solution. (https://dailymed.nlm.nih.gov/dailymed/fda/fdaDrugXsl.cfm?setid=4bd4d59c-eb3b-4a5e-9eb7-ae95b0a92bea&type=display
- [Background] Wang G, Peng X. A Review of Clinical Applications and Side Effects of Methotrexate in Ophthalmology. J Ophthalmol. 2020 Aug 11;2020:1537689. doi: 10.1155/2020/1537689. eCollection 2020. PMID 32850138
- [Background] Tables of Possible Side Effects for Commonly-Used Oncology Drugs. NIH. (https://ctep.cancer.gov/protocoldevelopment/sideeffects/drugs.htm